CLINICAL TRIAL: NCT00683189
Title: Effect of Warfarin in the Treatment of Metachromatic Leukodystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Mitra Assadi, M.D., Cooper University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP#07/063
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Metachromatic Leukodystrophy
Keywords: MLD
MeSH Terms: conditions — Leukodystrophy, Metachromatic | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Warfarin — Oral administration (QD), variable dosage: patients will undergo blood test for PT/INR at baseline and afterwards, at weekly bases for 4 weeks. The INR will be kept in a safe range of 2-2.5

SUMMARY:
Objectives/Purpose:

To determine the safety and efficacy of a Vitamin K (Vit K) antagonist (warfarin) in treating Metachromatic Leukodystrophy (MLD).

DETAILED DESCRIPTION:
Hypothesis:

Vit K has an essential role in biosynthesis of sulfatides and other sphingolopids in the brain. Administering warfarin, a Vit K antagonist, may ameliorate the phenotype in MLD by decreasing t he amount of sphingolipid storage in the neuronal cells.

Study Design Prospective: we will enroll eligible consenting subjects into the study. The study will not include a control group and the families and treating physicians are informed administration of the drug.

1. Duration of Treatment: 4 weeks
2. Pharmacological Intervention: The patients will receive warfarin 1.5 mg at the beginning of the study period. The dosage then will be adjusted to the INR values on weekly basis.
3. Clinical evaluation: The patients will undergo clinical assessment prior to starting the treatment and at the end of the treatment period. The clinical assessment will also include administration of Gross Motor Function Measure (GMFM), a clinical toll for evaluation of motor development in children.
4. Urine Sulfatide Quantification: Urine samples for quantification of the sulfatide level will be collected at the time of enrollment, after 2 weeks and at the end of treatment period.
5. Blood Monitoring: The patients will undergo blood test for PT/INR at baseline and afterwards, at weekly bases for 4 weeks. The INR will be kept in a safe range of 2-2.5. If the INR is greater than 4.0 the dosage of warfarin will be lowered and another blood draw will be performed in 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Children with MLD, 1 to 10 years of age who have received and failed bone marrow transplantation or are excluded from the treatment due to delayed diagnosis or any other reasons.

Exclusion Criteria:

* Any Children with MLD who are eligible for and might receive ABMT.
* Any Children with MLD who suffer with a bleeding disorder, moderate to severe anemia or any other hematological disorders.
* Any contraindications systemic for anti-coagulation

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Quantitative Neurological Assessment | 4 weeks
Urine Sulfatides Quantification | 4 weeks

SECONDARY OUTCOMES:
Brain MRI | before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paola Leone, Ph.D., Study Director — UMDNJ/SOM; Mitra Assadi, M.D., Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States